CLINICAL TRIAL: NCT01373931
Title: Effect of LY2216684 on Oral Contraceptive Pharmacokinetics in Healthy Female Subjects
Brief Title: A Study of LY2216684 in Healthy Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 12615; H9P-EW-LNCX (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-06-13; First posted 2011-06-15 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-03

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- OC + LY2216684 First, Then OC + Placebo (Experimental): 28-day lead-in period of Ortho Cyclen (OC; 28-day packet), followed by randomization to OC administered orally once daily for 28 days + 18 milligrams (mg) of LY2216684 administered concomitantly orally once daily for 21 days, followed by OC administered orally once daily for 28 days + placebo administered concomitantly orally once daily for 21 days.
  Interventions: Drug: LY2216684; Drug: Ortho Cyclen; Drug: Placebo
- OC + Placebo First, Then OC + LY2216684 (Experimental): 28-day lead-in period of OC (28-day packet), followed by randomization to OC administered orally once daily for 28 days + placebo administered concomitantly orally once daily for 21 days, followed by OC administered orally once daily for 28 days + 18 mg of LY2216684 administered concomitantly orally once daily for 21 days.
  Interventions: Drug: LY2216684; Drug: Ortho Cyclen; Drug: Placebo

INTERVENTIONS:
Drug: LY2216684 — Administered orally
Drug: Ortho Cyclen — 35 micrograms (mcg) ethinyl estradiol and 250 mcg norgestimate administered orally
Drug: Placebo — Administered orally

SUMMARY:
This study involves a single dose of 18 milligrams (mg) LY2216684 taken as 1 or 2 tablets by mouth. The study will evaluate effect of LY2216684 on the pharmacokinetics of an oral contraceptive Ortho Cyclen®. This study will run approximately 93 days.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy females, as determined by medical history and physical examination
* As it is possible that LY2216684 may cause the oral contraceptive tablet to be less effective than usual, participants will be required in addition to use double barrier methods of contraception from the Screening until 2 months after the post study follow-up. Additional barrier methods of contraception may include the following: a non-hormonal intrauterine device with spermicide; female condom with spermicide; contraceptive sponge with spermicide; diaphragm with spermicide; cervical cap with spermicide; a male sexual partner who agrees to use a male condom with spermicide; a sterile sexual partner; or abstinence (participants reporting abstinence who become sexually active while on the study must agree to use other additional barrier methods of contraception). The pregnancy test result must be negative at Screening and at each Check-in
* Have a body weight of >50 kilograms (kg)
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow for blood sampling as per the protocol
* Have normal blood pressure and pulse rate (sitting position) as determined by the investigator
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Lilly and the institutional review board (IRB) governing the site

Exclusion Criteria:

* Are currently enrolled in, have completed or discontinued within the last 30 days from, a clinical trial involving an investigational product other than the investigational product used in this study, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to Ortho Cyclen, LY2216684, or related compounds
* Are participants who have previously completed or withdrawn from this study or any other study investigating LY2216684 within 6 months prior to Screening
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Have a history or show evidence of significant active neuropsychiatric disease or have a history or suicide attempt or ideation
* Regular use of known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus infection (HIV) and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Are women with a positive pregnancy test or women who are lactating
* Intend to use over-the-counter or prescription medication (other than the acceptable oral contraceptive allowed in this study and influenza vaccinations) within 14 days prior to dosing unless deemed acceptable by the investigator and sponsor's medical monitor
* Have donated blood of more than 500 milliliter (mL) prior to lead-in phase Check-in (Day -1)
* Have an average weekly alcohol intake that exceeds 14 units per week, or are unwilling to stop alcohol consumption for 48 hours prior to each Check-in to the clinical research unit (CRU) [1 unit = 12 ounces (oz) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits]
* Consume 5 or more cups of coffee (or other beverages of comparable caffeine content) per day, on a habitual basis, or any participants unwilling to adhere to study caffeine restrictions
* Use of any tobacco- or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to the lead-in phase Check-in (Day -1) and during the study
* Have consumed grapefruit, starfruit, pomegranates, or products containing those items 7 days prior to enrollment or are unwilling to avoid them during the study
* Have a documented or suspected history of glaucoma
* Participants that have taken injectable contraceptives within 12 months of enrollment to this study or topical controlled delivery contraceptives (patch) for 3 months prior to enrollment into this study
* The history or presence of any contraindications to the combined oral contraceptive tablet including thrombosis and the history of any thromboembolic disease, recurrent jaundice, acute or chronic liver disease, migraines, undiagnosed vaginal bleeding, significant hyperlipidemia, and mammary, endometrial, or hepatic carcinoma (known or suspected)
* Participants determined to be unsuitable by the investigator for any reason

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomized, 2-period, 2-sequence crossover study with a lead-in period.
Groups:
- OC + LY2216684 / OC + Placebo: Lead-in Period: 28 days of Ortho Cyclen [OC; 21 days of 35 micrograms (mcg) ethinyl estradiol and 250 mcg norgestimate and 7 days of OC placebo]
  Period 1: OC + 18 milligrams (mg) of LY2216684 administered concomitantly orally, once daily for 21 days and 7 days of OC placebo
  Period 2: OC + LY2216684 placebo administered concomitantly orally, once daily for 21 days and 7 days of OC placebo
- OC + Placebo / OC + LY2216684: Lead-in Period: 28 days of OC (21 days of 35 mcg ethinyl estradiol and 250 mcg norgestimate and 7 days of OC placebo)
  Period 1: OC + LY2216684 placebo administered concomitantly orally, once daily for 21 days and 7 days of OC placebo
  Period 2: OC + 18 mg of LY2216684 administered concomitantly orally, once daily for 21 days and 7 days of OC placebo
Period: Lead-in Period
Arm/Group | OC + LY2216684 / OC + Placebo | OC + Placebo / OC + LY2216684
Started | 10 | 10
Received at Least 1 Dose of Study Drug | 8 | 10
Completed | 8 | 10
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0
Period: Period 1
Arm/Group | OC + LY2216684 / OC + Placebo | OC + Placebo / OC + LY2216684
Started | 8 | 10
Completed | 6 | 8
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2
Period: Period 2
Arm/Group | OC + LY2216684 / OC + Placebo | OC + Placebo / OC + LY2216684
Started | 6 | 8
Completed | 6 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | OC + LY2216684 / OC + Placebo | OC + Placebo / OC + LY2216684 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (8.9) | 30.7 (10.0) | 30.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 9 | 8 | 17
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax) of Ethinyl Estradiol and Norelgestromin
Description: The results presented are Geometric Least Squares (LS) mean. LS mean values were adjusted for treatment, sequence, period and participant.
Time Frame: Predose up to 24 hours post dose on Day 21
Population: All randomized participants who received at least 1 dose of study drug and had pharmacokinetics data to analyze Cmax. Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (90% Confidence Interval); unit: picograms/milliliter (pg/mL)
Groups:
- OC + LY2216684: Ortho Cyclen (OC) + 18 milligrams (mg) of LY2216684 administered concomitantly orally, once daily for 21 days and 7 days of OC placebo in both sequences
- OC + Placebo: OC + LY2216684 placebo administered concomitantly orally, once daily for 21 days and 7 days of OC placebo in both sequences
Arm/Group | OC + LY2216684 | OC + Placebo
Number analyzed (Participants) | 14 | 16
picograms/milliliter (pg/mL)
  Ethinyl Estradiol: number analyzed (Participants) | 14 | 15
  Ethinyl Estradiol | 79.0 [70.0 to 89.1] | 80.9 [71.8 to 91.2]
  Norelgestromin | 1438 [1301 to 1589] | 1574 [1427 to 1735]
Statistical Analysis 1: Comparison: OC + LY2216684 vs OC + Placebo; Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geometric LS mean is for ethinyl estradiol; Ratio of Geometric LS Mean = 0.976, 90% CI 2-sided [0.907 to 1.05]
Statistical Analysis 2: Comparison: OC + LY2216684 vs OC + Placebo; Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geometric LS mean is for norelgestromin; Ratio of Geometric LS Mean = 0.914, 90% CI 2-sided [0.842 to 0.991]

2. Primary Outcome: Pharmacokinetics: Time to Maximum Plasma Concentration (Tmax) of Ethinyl Estradiol and Norelgestromin
Time Frame: Predose up to 24 hours post dose on Day 21
Population: All randomized participants who received at least 1 dose of study drug and had pharmacokinetics data to analyze tmax. Participants were analyzed based on the treatment they received.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | OC + LY2216684 | OC + Placebo
Number analyzed (Participants) | 14 | 14
hour (h)
  Ethinyl Estradiol: number analyzed (Participants) | 13 | 13
  Ethinyl Estradiol | 2.00 [1.50 to 4.00] | 2.00 [1.50 to 4.00]
  Norelgestromin | 3.00 [1.50 to 4.00] | 2.03 [1.50 to 4.07]
Statistical Analysis 1: Comparison: OC + LY2216684 vs OC + Placebo; Test type: Superiority or Other; Wilcoxon Signed Rank Test; Median difference is for ethinyl estradiol; Median Difference (Final Values) = -0.25, 90% CI 2-sided [-0.73 to 0.51]
Statistical Analysis 2: Comparison: OC + LY2216684 vs OC + Placebo; Test type: Superiority or Other; Wilcoxon Signed Rank Test; Median difference is for norelgestromin; Median Difference (Final Values) = 0.00, 90% CI 2-sided [-0.50 to 0.50]

3. Primary Outcome: Area Under the Concentration-Time Curve Over a Dosing Interval (AUCτ) of Ethinyl Estradiol and Norelgestromin
Description: as for outcome 1
Time Frame: Predose up to 24 hours post dose on Day 21
Population: All randomized participants who received at least 1 dose of study drug and had pharmacokinetics data to analyze AUCτ. Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (90% Confidence Interval); unit: picograms*hour/milliliter (pg*hr/mL)
Arm/Group | OC + LY2216684 | OC + Placebo
Number analyzed (Participants) | 14 | 16
picograms*hour/milliliter (pg*hr/mL)
  Ethinyl Estradiol: number analyzed (Participants) | 14 | 14
  Ethinyl Estradiol | 888 [799 to 987] | 827 [744 to 918]
  Norelgestromin | 16156 [14626 to 17846] | 16079 [14575 to 17738]
Statistical Analysis 1: Comparison: OC + LY2216684 vs OC + Placebo; Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geometric LS mean is for ethinyl estradiol; Ratio of Geometric LS Mean = 1.07, 90% CI [1.00 to 1.15]
Statistical Analysis 2: Comparison: OC + LY2216684 vs OC + Placebo; Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geometric LS mean is for norelgestromin; Ratio of Geometric LS Mean = 1.00, 90% CI [0.944 to 1.07]

ADVERSE EVENTS:
Groups:
- OC Lead-in Period: Lead-in Period: 28 days of Ortho Cyclen [OC; 21 days of 35 micrograms (mcg) ethinyl estradiol and 250 mcg norgestimate and 7 days of OC placebo]
- OC + LY2216684: OC + 18 milligrams (mg) of LY2216684 administered concomitantly orally, once daily for 21 days and 7 days of OC placebo in both sequences
Arm/Group | OC Lead-in Period | OC + LY2216684 | OC + Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 12/18 | 13/16 | 13/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OC Lead-in Period (N=18) | OC + LY2216684 (N=16) | OC + Placebo (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 4 (4) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (4) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 6 (6) | 3 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 5 (5) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1) | 2 (2)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1) | 2 (2)
Vessel puncture site swelling (General disorders) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 7 (13) | 2 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 5 (7) | 3 (5)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (4) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Emotional poverty (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Panic reaction (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Piloerection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days